CLINICAL TRIAL: NCT07310745
Title: Low Dose Radiotherapy in Primary Indolent Cutaneous B-cell Lymphoma
Acronym: LDRT
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 263/2022/OSS/IRCCSRE
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Primary Indolent Cutaneous B-cell Lymphoma
Keywords: Primary indolent cutaneous B-cell Lymphoma; Low dose RT; Primary cutaneous marginal zone lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Primary indolent cutaneous B cell lymphomas (PCBCL) are rare: although data on outcomes and treatment are limited, traditionally they have been treated with radiation doses in excess of 24 Gy. Recently, some trials that patients with primary cutaneous indolent lymphoma managed with very low dose (4 Gy) RT (LDRT) have shown that high response rates and durable remission can be achieved; unfortunately, given the retrospective nature of these studies, the role of LDRT in indolent PMCL remains undefined. The objective of this retrospective multicentric trial is to investigate the efficacy of low-dose involved-field radiation therapy in patients with primary indolent cutaneous B-cell Lymphoma.

DETAILED DESCRIPTION:
Primary cutaneous B-cell lymphomas (PCBCL) represent approximately 20% of all primary cutaneous lymphoma and are defined by a restricted disease spread to the skin without evidence of extracutaneous involvement at diagnosis. They encompass three main types: primary cutaneous marginal zone lymphoma (PCMZL), primary cutaneous follicle center lymphoma (PCFCL) and primary cutaneous diffuse large B-cell lymphoma, leg type (PCDLBCL, LT), of which the first two entities are indolent. Radiotherapy (RT) is part of the therapeutic mosaic for PCBCL and recommended by both national and international guidelines for a localized disease pattern, conferring high local control rates with a conservative approach . Curative doses cover a range of 18-54 Gy and complete remission is common regardless of which treatment is used. There is accumulating evidence for a possible de-escalation of RT dose while maintaining high response rates and thereby opening a role for low-dose RT (LDRT), which has been successfully shown for other indolent non-Hodgkin lymphoma. However, the rarity of indolent PCBCL and retrospective nature of studies make a definitive dose recommendation troublesome.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Histological diagnosis of indolent B-cell lymphoma (follicular, marginal, NOS)
* Primary cutaneous location
* Early stage (I-II)
* First diagnosis or recurrence
* Low-dose radiotherapy treatment (4 Gy/2 sessions)

Exclusion Criteria:

* Aggressive histology lymphomas
* Advanced stages
* Extracutaneous localisation
* Radiotherapy dose administered > 4 Gy
* Patients without histological typing
* Patients without follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves adult patients with early-stage (I-II) primary cutaneous indolent B-cell lymphoma (PCBCL) treated with low-dose radiotherapy (4 Gy in two sessions). Patients with a confirmed histological diagnosis of indolent B-cell lymphoma (follicular, marginal, NOS) and adequate follow-up are included. Patients with aggressive lymphomas, advanced stages, extracutaneous localisations or radiotherapy doses greater than 4 Gy are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Local Progression-Free Interval in Irradiated Field | 12 months
  Time from the start of low dose radiotherapy (LDRT) to tumor progression within the irradiated field

SECONDARY OUTCOMES:
Acute toxicity | 4 weeks
  The occurence and severity of acute adverse events (toxicities)
Late toxicity | 12 weeks
  The occurrence and severity of late adverse events (toxicities)
Tumor response in irradated area | 12 weeks
  The response of the tumor in the irradiated area will be evaluated based on radiological imaging and/or clinical examination
Overall response rate (ORR) | 12 weeks
  The overall response rate is defined as the percentage of patients achieving a complete response (CR) or partial response (PR) in the irradiated sites, as assessed by the investigator using the Lugano classification criteria.
Overall survival (OS) | 24 months
  Overall Survival (OS) is defined as the time from the start of LDRT to the date of death from any cause.
Progression-Free Survival (PFS) | 24 months
  Progression-Free Survival (PFS) is defined as the time from the start of Low Dose Radiotherapy (LDRT) to the first observation of disease progression or relapse, or the date of the last follow-up if no progression is observed

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL IRCCS di Reggio Emilia - Sc Radioterapia, Reggio Emilia, Italy

REFERENCES:
- [Background] Christensen L, Cooper K, Honda K, Mansur D. Relapse rates in patients with unilesional primary cutaneous B-cell lymphoma treated with radiation therapy: a single-institution experience. Br J Dermatol. 2018 Nov;179(5):1172-1173. doi: 10.1111/bjd.16783. Epub 2018 Jul 27. No abstract available. PMID 29761874
- [Background] Senff NJ, Noordijk EM, Kim YH, Bagot M, Berti E, Cerroni L, Dummer R, Duvic M, Hoppe RT, Pimpinelli N, Rosen ST, Vermeer MH, Whittaker S, Willemze R; European Organization for Research and Treatment of Cancer; International Society for Cutaneous Lymphoma. European Organization for Research and Treatment of Cancer and International Society for Cutaneous Lymphoma consensus recommendations for the management of cutaneous B-cell lymphomas. Blood. 2008 Sep 1;112(5):1600-9. doi: 10.1182/blood-2008-04-152850. Epub 2008 Jun 20. PMID 18567836
- [Background] Willemze R, Cerroni L, Kempf W, et al. The 2018 update of the WHO-EORTC classification for primary cutaneous lymphomas. Blood. 2019;133(16):1703-1714. Blood. 2019 Sep 26;134(13):1112. doi: 10.1182/blood.2019002852. No abstract available. PMID 31558559
- [Background] Willemze R, Hodak E, Zinzani PL, Specht L, Ladetto M; ESMO Guidelines Committee. Primary cutaneous lymphomas: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv30-iv40. doi: 10.1093/annonc/mdy133. No abstract available. PMID 29878045
- [Background] Nicolay JP, Wobser M. Cutaneous B-cell lymphomas - pathogenesis, diagnostic workup, and therapy. J Dtsch Dermatol Ges. 2016 Dec;14(12):1207-1224. doi: 10.1111/ddg.13164. PMID 27992127
- [Background] Dippel E, Assaf C, Becker JC, von Bergwelt-Baildon M, Beyer M, Cozzio A, Eich HT, Follmann M, Grabbe S, Hillen U, Klapper W, Klemke CD, Lamos C, Loquai C, Meiss F, Mestel D, Nashan D, Nicolay JP, Oschlies I, Schlaak M, Stoll C, Vag T, Weichenthal M, Wobser M, Stadler R. S2k Guidelines - Cutaneous Lymphomas Update 2016 - Part 1: Classification and Diagnosis (ICD10 C82 - C86). J Dtsch Dermatol Ges. 2017 Dec;15(12):1266-1273. doi: 10.1111/ddg.13372. Epub 2017 Nov 28. No abstract available. PMID 29193659